CLINICAL TRIAL: NCT03755661
Title: Alcohol and Implicit Process in Sexual Risk Behavior in MSM Supplement
Brief Title: MI With Text Messaging to Reduce Sexual Risk and Hazardous Drinking Among MSM
Acronym: MI&TXT4MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Tibor Palfai, Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3468a; 3R01AA022301-02S1 (NIH)
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-03

CONDITIONS: Alcohol; Harmful Use; Sex, Unsafe
MeSH Terms: conditions — Unsafe Sex

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is not provided with randomization information for the subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This intervention arm is a combined in-person text messaging intervention
  Interventions: Behavioral: MI&TXT4MSM
- Assessment Only Control (No Intervention): The is the assessment only comparison condition

INTERVENTIONS:
Behavioral: MI&TXT4MSM — brief in-person intervention followed by text messaging
  Arms: Intervention

SUMMARY:
This is a small pilot study to provide effect size estimates for a brief intervention designed to reduce hazardous drinking and sexual risk behavior among men who have sex with men. The intervention consists of an "in-person" brief motivational intervention followed by a series of text messages related to alcohol and sexual risk reduction. The primary outcome is heavy drinking episodes and frequency of condomless anal intercourse at 3 months.

DETAILED DESCRIPTION:
This is a pilot study designed to provide initial effect size estimates for an intervention addressing hazardous drinking and sexual risk behavior among men who have sex with men. In this study, 24 participants initially recruited through advertisements in the community will be randomly assigned to either Assessment Only or Intervention Condition. Those in the Assessment Only condition will complete baseline, 6-week, 3-month and 6-month assessments. Those in the intervention condition will receive a 50-min brief intervention in person followed by 6 weeks of tailored app-based messaging to support the intervention content, then another 6-weeks of goal setting text-based messages. Data will be analyzed to determine effect sizes of the intervention on key alcohol use and sex risk outcomes. The primary outcome will be 3-month outcomes, controlling for corresponding baseline outcomes.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 heavy drinking episode or consumption of more than 14 drinks per week over the past month
* At least 1 condomless anal sex episode in past 3 months
* Score of 3 or greater on the Kinsey Scale (Kinsey et al., 1948) indicating at least "equally heterosexual and homosexual". Scale ranges from 0 (exclusively heterosexual) to 6 (exclusively homosexual)

Exclusion Criteria:

* Alcohol treatment currently or in past 3 years
* Bipolar disorder or schizophrenia treatment
* Exclusive monogamous relationship

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — identify as male
Enrollment: 24 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University Department of Psychological and Brain Science, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared following release within one year of the trial end to investigators who make specific requests in writing regarding analysis plans. Plans will be reviewed with co-investigators to ensure that there is no overlap with planned analyses. Specific de-identified data set will be provided to other researchers after this review
Time Frame: Data will be available one year after the trial end. They will be available for investigators to request up to 5 years following their release
Access Criteria: Researcher with specified analytic request.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through social media ads and the study was conducted at a university laboratory that is affiliated with a psychological services clinic
Pre-assignment Details: Eligibility was confirmed at the in-person session. Randomization occurred following baseline assessment
Groups:
- Assessment Only Control: This condition includes only assessment measures. It is used as the comparison condition to the intervention under study.
Period: Overall Study
Arm/Group | Intervention | Assessment Only Control
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Assessment Only Control | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.18 (7.26) | 30.75 (7.79) | 30.48 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 9 | 20
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Heavy Drinking Episodes NIAAA Criteria (5 or More Drinks on a Single Occasion)
Description: Number of heavy drinking episodes in the past 30 days. This question is an open ended question that asks the participant to report the number of times in the past 30 days that he has consumed 5 or more drinks on a single occasion [no scale]. Higher score is a worse outcome, range 0-30
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: heavy drinking episodes
Arm/Group | Intervention | Assessment Only Control
Number analyzed (Participants) | 11 | 12
heavy drinking episodes | 3.09 (3.62) | 5.33 (3.42)
Statistical Analysis 1: Comparison: Intervention vs Assessment Only Control; pilot study to calculate effect size, study is not powered to detect significant group differences; Test type: Other — pilot data to estimate effect size f-squared as the parameter as primary outcome; p = .048, Regression, Linear — provide inferential statistics for data completion. Study is not designed to detect significant differences between groups; R-square change = .12; F-change (1, 20) = 4.44; Computed f-squared as effect size estimate where baseline value of heavy drinking episodes entered in step 1 and condition in step 2 f- squared = .22

2. Primary Outcome: Number of Condomless Anal Intercourse Episodes (CAI) From the Sexual Behaviors Survey (Gordon et al., 2007) is Used to Measure Sexual Risk [Main Time Point at 3 Month Follow-up]
Description: Frequency of CAI in past 90 days. This is an open ended question where the Participant report the frequency of condomless anal intercourse episodes over a period of 90 days [no scale] Range from 0-90
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: condomless anal intercourse episodes
Arm/Group | Intervention | Assessment Only Control
Number analyzed (Participants) | 11 | 12
condomless anal intercourse episodes | 1.54 (2.46) | 4.33 (6.12)
Statistical Analysis 1: Comparison: Intervention vs Assessment Only Control; pilot trial to compute effect size estimate; Test type: Superiority — The main outcome variable is f-squared as an estimate of differences between conditions controlling for baseline value. A statistical test is provided only for completeness as this study is not powered to detect significant effects; p = .34, Regression, Linear — F-change (1, 20) = 0.97; Computed f-squared as effect size estimate where baseline value of CAI entered in step 1 and condition in step 2 f- squared = .05, r-squared change = .04

3. Primary Outcome: Modified Daily Drinking Questionnaire- Typical Number of Standard Drinks Per Week Over the Past Month
Description: Average quantity of alcohol use per week in the past 30 days. Participants complete a seven day calendar which reflects the typical number of standard drinks that they have consumed for each day of the week over the past 30 days. The number of drinks can range from 0 to an unlimited high number. A higher number of drinks listed in the week is reflective of a worse outcome
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Average number of drinks per week
Arm/Group | Intervention | Assessment Only Control
Number analyzed (Participants) | 11 | 12
Average number of drinks per week | 9.45 (6.57) | 11.58 (6.14)
Statistical Analysis 1: Comparison: Intervention vs Assessment Only Control; Test type: Superiority — This is a pilot trial to estimate effect sizes and not powered to detect significant differences; p = .20, Regression, Linear — data provided for completeness, not powered to test differences; F-change (1, 20) = 1.80; Computed f-squared as effect size estimate where baseline value of CAI entered in step 1 and condition in step 2 f- squared = .09, r-squared change = .058

4. Secondary Outcome: Young Adult Alcohol Consequences Questionnaire [Alcohol]
Description: Number of alcohol-related consequences in the past month. This is the 48-item Yes/No version of the YAACQ. The range for the score is 0-48. Higher score is a worse outcome
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Assessment Only Control
Number analyzed (Participants) | 11 | 12
score on a scale | 6.45 (6.62) | 9.41 (7.41)
Statistical Analysis 1: Comparison: Intervention vs Assessment Only Control; Pilot trial not powered to detect significant group differences; Test type: Superiority — Pilot trial not powered to detect significant group differences. Data from analyses presented for completeness. Primary outcome is effect size estimates; p = .19, Regression, Linear; F-change (1, 20) = 1.83; Computed f-squared as effect size estimate where baseline value of CAI entered in step 1 and condition in step 2 f- squared = .09, r-squared change = .048

5. Other Pre Specified Outcome: Number of CAI Past 6 Weeks From the Sexual Behaviors Survey Item Described Above.
Description: The number of condomless anal intercourse episodes (CAI) in the 6 weeks following the baseline as an additional outcome
Time Frame: 6 -weeks
Measure: Mean (Standard Deviation); unit: condomless anal intercourse episodes
Arm/Group | Intervention | Assessment Only Control
Number analyzed (Participants) | 11 | 11
condomless anal intercourse episodes | 0.91 (0.94) | 1.63 (1.56)
Statistical Analysis 1: Comparison: Intervention vs Assessment Only Control; Not powered to test significant differences. provide data on effect size estimate below; Test type: Superiority; p = .26, Regression, Linear — F-change (1, 19) = 1.34; [other analysis details as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to the 6 month outcome following enrollment. This corresponds to the time period from initial enrollment to study completion
Groups:
- Intervention: This intervention arm is a combined in-person text messaging intervention
  MI&TXT4MSM: brief in-person intervention followed by text messaging
  No adverse events
- Assessment Only Control: The is the assessment only comparison condition
  No adverse events
Arm/Group | Intervention | Assessment Only Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT03755661/Prot_SAP_000.pdf